CLINICAL TRIAL: NCT07317167
Title: Evaluating a Water Safety Plan Intervention in Ghana
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Aquaya Institute (Other)
Collaborators: Kwame Nkrumah University of Science and Technology (KNUST) (Unknown); Conrad N. Hilton Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WSP Evaluation
Record Dates: First submitted 2025-11-20; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Water Quality; Water Treatment; Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water Safety Plan Intervention Arm (Experimental): Water Safety Plans
  Interventions: Other: Water Safety Plans
- Control Arm (No Intervention): No Water Safety Plans: Water systems will continue to manage their water supplies without the introduction of water safety plans.

INTERVENTIONS:
Other: Water Safety Plans — Water safety plans will be implemented at the water system level as a holistic tool for ensuring the safety of drinking water supplies from source to tap. World Health Organization guidance will be followed for implementation and recommended water safety planning steps will be followed such as assembling a WSP Team, describing the water supply, hazard identification and risk assessment, developing and implementing an incremental improvement plan, monitoring control measures to verify the effectiveness of the WSP, and continuously documenting, reviewing, and improving WSP implementation.
  Arms: Water Safety Plan Intervention Arm

SUMMARY:
The objective of this study is to evaluate the effects of water safety plans (WSPs) in rural Ghana. The investigators aim to evaluate the effects of WSPs on water supply system infrastructure, water availability and reliability, water quality, consumer perceptions, water service provider management and financial sustainability, climate resilience, equity, and consumer health.

DETAILED DESCRIPTION:
Much of the global population is exposed to contaminated drinking water. In piped systems, it is often easier to mitigate at the water supplier level where it can be centrally managed. A water safety plan (WSP) is a holistic tool for proactively ensuring the safety of drinking water supplies from source to tap, and the World Health Organization (WHO) recommends this systematic risk assessment and preventive management approach for water systems.

While application of WSPs has spread, systematic evidence for their implementation and effectiveness in improving water quality and health is limited, particularly in low-resource settings.

The objective of this study is to evaluate the impact of WSPs on water supply system infrastructure, water availability and reliability, water quality, consumer perceptions, water service provider management and financial sustainability, climate resilience, equity, and consumer health. The investigators will use a randomized controlled trial across 92 piped water supply systems serving small towns and rural areas in Ghana to test the effectiveness of WSPs. The investigators will collect data at baseline before the intervention is implemented, and at endline approximately 2 years after implementation begins. The investigators will also conduct a process evaluation of the WSP implementation quality.

ELIGIBILITY:
Eligibility to receive the intervention was determined by water system criteria:

Inclusion Criteria:

* Water systems must be operated by a partnering private, non-profit water supplier.
* Water systems must be functional during baseline data collection.

To be eligible to participate in household surveys or focus group discussions, participants need to be at least 18 years of age and a customer of a eligible water system. To be eligible to participate in health care facility interviews, participants must be at least 18 years of age and work at a health care facility that serves community members using the included water system.

Exclusion Criteria:

* Water systems did not meet both of the above inclusion criteria.
* Water systems had already implemented a water safety plan.
* Water systems were involved in another ongoing research trial with similar expected outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Free chlorine residue in water at point of collection (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Free chlorine residue in water at point of collection (public standpipes and private taps) at or above target level of 0.2 mg/L, and at or above detectable level of 0.1 mg/L
E. coli in water at point of collection (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  E. coli in water at point of collection (binary and categorical)
Total coliform in water at point of collection (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Total coliform in water at point of collection (binary)
Turbidity of water at point of collection (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Turbidity measured in NTU in water at point of collection
Reliability/availability of water (water supply impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Reliability/availability of water based on (1) service provider documented interruptions, and (2) consumer reported service interruptions

SECONDARY OUTCOMES:
Consumer satisfaction (consumer perception impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Household respondent satisfaction with water supplier. They will be considered satisfied if they report they are either satisfied or very satisfied with the water supplier. They will be considered dissatisfied if they report they are either dissatisfied or very dissatisfied with the water supplier.
Household use of enrolled piped water system for drinking (consumer perception impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Household use of enrolled piped water system for drinking (binary).
Households perceive water quality issues with piped water system (consumer perception impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Household respondents report water quality issues with the taste, odor, or appearance of supplied water.
Number of complaints (consumer perception impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Number of complaints regarding the service or quality of water. This will be measured based on (1) household self-reporting, and (2) water system reports or records.
Prevalence of diarrhea (health impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Prevalence of reported diarrhea in the past two weeks. Diarrhea is defined as 3 or more loose or watery stools within 24 hours. Measured for a household's youngest child <5 years old, and any household member showing symptoms.
Blood in stool (health impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Prevalence of reported blood in stool in the past two weeks. Measured for a household's youngest child <5 years old, and any household member showing symptoms.
Prevalence of severe diarrhea (health impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Prevalence of reported severe diarrhea in the past two weeks. Defined as having a fever and either diarrhea or blood in stool. Measured for a household's youngest child <5 years old.
Prevalence of acute respiratory infection (health impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Prevalence of reported severe or non-severe acute respiratory infection (ARI) in the past two weeks. A severe ARI is defined as having a fever and either a cough or difficulty breathing. A non-severe ARI is defined as having a cough or difficulty breathing. Measured for a household's youngest child <5 years old.
Number of clinic visits for water-related illness (health impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Clinical visits will be assessed based on (1) the number of clinic visits reported by households for diarrhea-related illness, and (2) records for the number of cases of water-related illness in patients who visited healthcare facilities serving the included communities.
E. coli in stored water at point of consumption (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  E. coli in stored household water at point of consumption (binary and categorical)
Total coliform in stored water at point of consumption (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Total coliform in stored household water at point of consumption (binary)
Free chlorine residue in stored water at point of consumption (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Free chlorine residue in stored household water at point of consumption at or above target level of 0.2 mg/L, and at or above detectable level of 0.1 mg/L
Total chlorine residue in stored water at point of consumption (water quality impacts) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Total chlorine residue in stored household water at point of consumption at or above target level of 0.2 mg/L, and at or above detectable level of 0.1 mg/L

OTHER OUTCOMES:
Number of risk factors identified by sanitary inspections (operational outcomes) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Number of risk factors identified by sanitary inspections of water system infrastructure including the water source, water tank, distribution system, and standpipes.
Quality and use of written documentation for water system management (operational outcomes) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Quality and use of written documentation for water system management including an operational monitoring plan, compliance monitoring plan, standard operating procedures, troubleshooting manual, maintenance schedule, and operator training program. It will be assessed whether written documentation exists, and if yes, whether it is detailed or incomplete and lacking detail. Water operators will also report if the written procedures are fully implemented in practice or not. This is intended to evaluate the professionalization and management of the water systems.
Cost recovery (financial outcomes) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Financial sustainability/cost recovery (ratio of revenue collected to operating costs) of the system
Number of meetings (institutional outcomes) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  (1) Number of internal and external water safety meetings, and (2) Number of consumer water safety training or awareness events
Documentation of climate related risks and response (climate resilience outcomes) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Documentation of climate related risks and response including whether climate-related information for the water supply system has been identified and documented, climate-related hazards related to events like heavy rainfall, flooding, and drought have been identified and prioritized, and an emergency response plan has been prepared. It will be assessed whether each aspect has been completed, and if yes whether it has been partially undertaken, but not documented; or fully undertaken and documented.
Identification and prioritization of disadvantaged groups by the water supplier (equity outcomes) | Baseline (before intervention), Endline (approximately 24-months after the start of the intervention)
  Identification of disadvantaged groups in the water service area has been completed by the water supplier and they have been prioritized for participation or the service provider has made improvements to the water system to address inequalities between disadvantaged and non-disadvantaged groups. It will be assessed whether each aspect has been completed, and if yes whether it has been partially undertaken, but not documented; or fully undertaken and documented.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Bauza, Principal Investigator — The Aquaya Institute
Locations (1):
- The Aquaya Institute, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available.